CLINICAL TRIAL: NCT04531254
Title: Understanding the Impact of Public Health Measures Planned for School Reopening During COVID-19 Using Simulation Exercises
Brief Title: Back to School COVID-19 Simulation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Michelle Science, Infectious Disease Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1000071861
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Covid19; Schools
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Masking at all times (Experimental): Children in this group will be asked to wear a face mask/covering in the classroom and common areas during the simulation
  Interventions: Behavioral: Wearing a face mask at all times
- No mask/masking when physical distancing is not maintained (No Intervention): Children in this group will not be asked to wear a mask (JK-Grade 4) or only asked to wear a mask when physical distancing in the classroom cannot be maintained (Grade 5-Grade 12) during the simulation

INTERVENTIONS:
Behavioral: Wearing a face mask at all times — Children in this group will be asked to wear a face mask in the classroom and common areas during the simulation
  Arms: Masking at all times

SUMMARY:
This will be a prospective study simulating return to school for two full days prior to the start of the school year in September. Volunteer students and teachers from six grade ranges will be recruited to participate in the study. In each grade range, there will be two classes that will participate, one that will be assigned to wear face masks/coverings at all times (experimental group/class) and the other that will not wear face masks/coverings at all times (control group/class). Students will be randomized to either the masking at all times (experimental across all grades) or no masking (control across JK-Grade 4) / masking only when physical distance can be maintained (control across Grade 5-Grade 12) class in their appropriate grade. Personal behaviours and person-to-person interactions will be recorded using video cameras. In addition, a safe biological indicator will be applied to the hands to simulate potential asymptomatic infection in a subset of students. Other students will have sanitizer applied so that students are blinded to who has the indicator. Cameras will be used to document how the indicator moves throughout the classroom.

DETAILED DESCRIPTION:
Grade ranges will include 1) Senior Kindergarten (children who have just completed JK or SK in the 2019-2020 year), 2) Grades 1-2, 3) Grades 3-4, 4) Grades 5-6, 5) Grades 7-8 and 6) high school. A total of 14 teachers and up to 240 students will be recruited. Final class sizes will be in accordance with Ministry of Education and public health guidelines.

ELIGIBILITY:
Inclusion Criteria:

• To be included in the study, students must have attended a structure learning environment during 2019-2020 school year and provide informed consent (student in Grade 7 or older) or parental consent (SK - Grade 6) and assent (if appropriate). To be included in the study, teachers must be certified teachers and provide informed consent to participate.

Exclusion Criteria:

* require additional resources or support beyond what can be provided by the single class teacher
* have been exposed to an individual that has tested positive for COVID-19 in the 14 days prior to the simulation
* test positive for COVID-19 in the 14 days prior to the simulation
* have signs or symptoms of COVID-19, as identified on the screening form (See Screening Form) before the simulations
* travel outside Canada in the last 14 days
* known hypersensitivity or allergy to the biological indicator (Fluorescein dye/GloGerm)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 174 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Total number of hand-to-face contacts per participant per hour | Day 2
  The number of touches to the face made per hour in the simulated school environment

SECONDARY OUTCOMES:
Total number of hand-to-mucus membrane contacts per participant per hour | Day 2
  The number of touches to the eyes, nose, mouth made per hour in the simulated school environment
Total number of hand-to-non-mucus membrane contacts per participant per hour | Day 2
  The number of touches to the skin (not eyes, nose, mouth) made per hour in the simulated school environment
Total number of instances where participants are within 1 and 2 meters of each other | Day 2
  The number of instances where 1 and 2 meter distance between participants is breached in the classroom
Total number of glo germ transfers to another person | Day 2
  The number of children within a classroom with Glo Germ on the hands/face
Total number of glo germ transfers to teacher | Day 2
  The presence of Glo Germ on the hands/face of teacher within the same classroom
Total number of glo germ transfers to a surface | Day 2
  The number of surfaces in the classroom with Glo Germ
Total number of instances of hand holding per participant per hour | Day 2
  The count of hand holding instances with another person per hour in the simulated school environment
Total number of touches to another person per participant per hour | Day 2
  The count of touches to another person per hour in the simulated school environment
Total number of hand hygiene actions per participant per hour | Day 2
  The count of hand hygiene actions (i.e., hand washing, hand sanitizer) per participant per hour
Total number of mask removals per participant per hour | Day 2
  The number of times a participant in a masking group removes their mask per hour in the simulated school environment
Teacher concerns measured using study-specific post-simulation questionnaire | Day 2
  A study specific questionnaire that examines teacher anxiety and mental health
Teacher concerns measured using semi-structured group interviews | Day 2
  A study specific semi-structured interview examining the factors throughout the day (hand hygiene, mask use, physical distancing) that impacted the teaching experience
Student concerns measured using study-specific post-simulation questionnaire | Day 2
  A study specific questionnaire that examines student anxiety and mental health
Student concerns measured using semi-structured group interviews | Day 2
  A study specific semi-structured interview examining the factors throughout the day (hand hygiene, mask use, physical distancing) that impacted the learning experience
Identify activity types that influence touching behaviour | Day 2
  The count of each type of activity participants are engaged in while touching others or surfaces in the simulated school environment

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Science, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Science M, Caldeira-Kulbakas M, Parekh RS, Maguire BR, Carroll S, Anthony SJ, Bitnun A, Bourns LE, Campbell DM, Cohen E, Dodds A, Dubey V, Friedman JN, Greenwood JL, Hopkins JP, Imgrund R, Korczak DJ, Looi T, Louca E, Mertz D, Nashid J, Panzera G, Schneiderman JE, Schwartz KL, Streitenberger L, Vuppal S, Walsh CM, Juni P, Matava CT; Back-to-School COVID-19 School Study Group. Effect of Wearing a Face Mask on Hand-to-Face Contact by Children in a Simulated School Environment: The Back-to-School COVID-19 Simulation Randomized Clinical Trial. JAMA Pediatr. 2022 Dec 1;176(12):1169-1175. doi: 10.1001/jamapediatrics.2022.3833. PMID 36279142